CLINICAL TRIAL: NCT03987906
Title: Symptom Screening With Targeted Early Palliative Care (STEP) Versus Usual Care for Patients With Advanced Cancer: A Randomized Controlled Trial
Brief Title: Symptom Screening With Targeted Early Palliative Care (STEP) Versus Usual Care for Patients With Advanced Cancer
Acronym: STEP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 pandemic
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Kingston Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-5007
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Cancer
Keywords: Palliative Care; Symptom control; Quality of life; Satisfaction with care; Targeted referral; Randomized controlled trial
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Symptom screening with Targeted Early Palliative Care (STEP) (Experimental): The experimental arm receives routine symptom screening at every outpatient visit; if symptoms are above a certain threshold, then a triggered email is sent to a triage nurse, who calls the patient to offer early referral to and follow-up by a symptom control and palliative care team.
  Interventions: Behavioral: Symptom screening with Targeted Early Palliative Care (STEP)
- Standard Oncology Care (No Intervention): The control arm receives standard oncology care, which includes routine symptom screening at every outpatient visit.

INTERVENTIONS:
Behavioral: Symptom screening with Targeted Early Palliative Care (STEP) — The experimental arm receives routine symptom screening at every outpatient visit; if symptoms are above a certain threshold, then a triggered email is sent to a triage nurse, who calls the patient to offer early referral to and follow-up by a symptom control and palliative care team.
  Other Names: STEP
  Arms: Symptom screening with Targeted Early Palliative Care (STEP)

SUMMARY:
Palliative care is defined as multidisciplinary care that increases quality of life (QOL) for patients with a life-threatening illness. Although it is known that patients with the most severe physical and psychological symptoms have the greatest need for palliative care, these patients are often not referred to palliative care services in a timely manner.

The investigators have developed a system called STEP (Symptom screening with Targeted Early Palliative care) that identifies patients with high symptom burden in order to offer them timely access to palliative care. The investigators are conducting a multi-center trial at Princess Margaret Cancer Centre and Kingston General Hospital to compare STEP with usual symptom screening in medical oncology clinics.

DETAILED DESCRIPTION:
Randomized controlled trials have shown that when patients with advanced cancer were referred early to specialized palliative care teams, they had improved QOL, symptom control, and greater satisfaction with their cancer care. Such routine specialized palliative care intervention, while effective, may be challenging to enact broadly with widespread shortages of palliative care physicians. STEP systematically identifies patients with the greatest need, using symptom screening at every outpatient visit, with triage and targeted referral to palliative care. This could reduce resource use while directing care to the most vulnerable.

Consenting patients from Breast, Lung, Gastrointestinal, Genitourinary, and Gynecology medical oncology clinics will be assigned randomly either to receive STEP or to follow usual symptom screening. All patients will complete questionnaires measuring outcomes of QOL, symptom control, depression, and satisfaction with care at recruitment, 2, 4 and 6 months. The investigators will measure the impact of STEP on these outcomes, compared to screening alone.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of stage IV cancer (advanced); hormone-refractory for breast or prostate cancer; stage III or IV for lung cancer and pancreatic cancer; patients with stage III cancer and poor clinical prognosis, e.g. ovarian or esophageal cancer, will be included at the discretion of the oncologist
* ECOG performance status ≤ 2 (estimated by primary oncologist)
* Prognosis of 6-36 months (estimated by primary oncologist)
* Patient completes symptom screening in outpatient clinic electronically

Exclusion Criteria:

* Insufficient English literacy to complete questionnaires
* Inability of pass the cognitive screening test (SOMC - Short Orientation Memory Concentration test score <20 or >10 errors)
* Receiving specialized palliative care within the last 6 months prior to screening, per chart and patient statement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Patient Heath Related Quality of Life (HRQL) as measured by the FACT-G7. | 6 months after enrollment.
  The FACT-G7 (Functional Assessment of Cancer Therapy-General 7 item) is a 7-item measure for quality of life that has been validated in patients with advanced cancer. Total score ranges from 0-28, higher scores indicate better quality of life.

SECONDARY OUTCOMES:
Patient Heath Related Quality of Life (HRQL) as measured by the FACT-G7. | 2 and 4 months after enrollment
  The FACT-G7 (Functional Assessment of Cancer Therapy-General 7 item) is a 7-item measure for quality of life that has been validated in patients with advanced cancer. Total score ranges from 0-28, higher scores indicate better quality of life.
Symptom control | 2, 4 and 6 months after enrollment
  Symptom control is measured by the 11-item ESAS-r-CS (Edmonton Symptom Assessment System-revised plus constipation and trouble sleeping). ESAS total distress score ranges from 0-110, higher scores indicate worse symptom burden.
Depression | 2, 4, and 6 months after enrollment
  Depression is measured by the Patient Health Questionnaire (PHQ-9). Total score ranges from 0-27, higher scores indicate worse depression.
Patient satisfaction with care. | 2, 4, and 6 months after enrollment
  Satisfaction with care is measured by the FAMCARE-P16 (Family Satisfaction with Cancer Scale modified for patients). Total score ranges from 16-80, higher scores indicate greater satisfaction with care.

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Zimmermann, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - Kingston General Hospital, Kingston, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No